CLINICAL TRIAL: NCT06185816
Title: Non-Invasive Pulsed Radiofrequency for the Treatment of Neuropathic Pain
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Hah, Associate Professor, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 71629
Record Dates: First submitted 2023-12-16; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Pain, Nerve
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Treatment (Active Comparator): ACTIVE treatment will be conducted by the study PIs, who are licensed pain physicians, Participants will receive 3 treatments, once weekly, for three weeks. Treatments are about 20 minutes long. The Stimpod being used is FDA cleared and is commercially available.
  The treatment is a non-invasive pulsed radio frequency current that emits a high frequency magnetic field. It has a pulse width of 0.2ms, a pulse rate of 2Hz and an intensity between 0 - 30ma. There is a 'beep' sound as the pulses occur. There are 2 electrodes used - one is the indifferent electrode that is placed on the skin at a suitable distance away from the active electrode and the other, an active electrode - is a probe that is applied to the target nerve to treat the mononeuropathy
  Interventions: Device: Active Treatment
- Non-Active Treatment (Sham Comparator): Participants enrolled in the non-active arm will receive 3 treatments, once weekly, for three weeks. After the trial is completed, participants will be offered three free treatments.
  The placebo device will be inert with nil current emitted however the device will look and be used in exactly the same way. There will also be a 'beep' sound emitted and only the investigator will know the difference. The placebo device will not deliver any electrical stimulation.
  Interventions: Device: Non-active Treatment

INTERVENTIONS:
Device: Active Treatment — The treatment is a non-invasive pulsed radio frequency current that emits a high frequency magnetic field. It has a pulse width of 0.2ms, a pulse rate of 2Hz and an intensity between 0 - 30ma. There is a 'beep' sound as the pulses occur. There are 2 electrodes used - one is the indifferent electrode that is placed on the skin at a suitable distance away from the active electrode and the other, an active electrode - is a probe that is applied to the target nerve to treat the mononeuropathy
  Arms: Active Treatment
Device: Non-active Treatment — The placebo device will be inert with nil current emitted however the device will look and be used in exactly the same way. There will also be a 'beep' sound emitted and only the investigator will know the difference. The placebo device will not deliver any electrical stimulation.
  Arms: Non-Active Treatment

SUMMARY:
The purpose of this study is to examine non-invasive pulsed radiofrequency (NIPRF) and the effect it has on chronic neuropathic pain. Chronic neuropathic pain after peripheral nerve injury most often occurs in the context of post-traumatic or post-surgical pain. It is often treated with nerve blocks, prescription medication, physical therapy, neuromodulation, and surgery. The study team will be examining the efficacy of NIPRF and determining if it would be an appropriate treatment for chronic neuropathic pain after peripheral nerve injury.The Stimpod used in the present study is FDA approved and will be used for on label purposes.

ELIGIBILITY:
Inclusion Criteria:

* -Adults aged 18 or older with clinically diagnosed chronic neuropathic pain after peripheral injury defined as persistent or recurrent neuropathic pain caused by a peripheral nerve lesion, history of a plausible nerve trauma, pain onset in temporal relation to the trauma, and pain distribution within the innervation territory of a peripheral nerve (or nerves). Negative and positive sensory symptoms or signs must be compatible with the innervation territory of the affected nerve. Can be posttraumatic, post-surgical, nerve compression, nerve ischemia with or without loss of motor function
* Positive response (at least 50% pain relief) to diagnostic nerve block at the suspected site of CNP-PI.
* Continued pain despite conservative therapy for a minimum of 12 weeks
* Stable dosage of analgesic medications for at least 30 days, and willingness to refrain from trialing new analgesic medications for three weeks after randomization
* Worst pain intensity of ≥5/10 on the Numeric Rating Scale (NRS) of Pain (0-10) at the CNP-PI site at enrollment
* English-speaking
* Ability and willingness to complete online and phone assessments

Exclusion Criteria:

* Conditions causing inability to complete assessments (education, cognitive ability, mental status, medical status)
* Cancer diagnosis, active malignant neoplasm (metastatic or local) or evidence of paraneoplastic syndrome
* Painful polyneuropathy (e.g., metabolic, autoimmune, familial, infectious disease, environmental toxins, treatment with neurotoxic drug)
* Chronic central neuropathic pain (e.g., spinal cord injury, brain injury, multiple sclerosis)
* Peripheral vascular disease
* Diabetic neuropathy
* Other active implantable devices (e.g., implantable cardioverter defibrillator, spinal cord stimulator, dorsal root ganglion stimulator, sacral nerve stimulator, deep brain stimulator, intrathecal pump)
* Pregnancy, breastfeeding, or planning to conceive
* Systemic infection or local infection at the anticipated NIPRF treatment sites
* Interventional procedure and/or surgery to treat CNP-PI in the last 30 days (subjects should be enrolled 30 days after last procedure, for prior ablative treatment must be enrolled at least 3 months after last procedure)
* Epilepsy
* Metal implants within the target treatment area of the NIPRF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Response Rate | After Three Weeks of Starting Treatment